CLINICAL TRIAL: NCT07210931
Title: A Cluster Randomized Trial in Patients With Knee Osteoarthritis Comparing Self-Managed Exercise in Fitness Centers With Physiotherapist-Supervised Exercise in Primary Care
Brief Title: Self-managed vs Supervised Exercise for Knee OA
Acronym: SELFIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marius Henriksen (Other)
Collaborators: University of Copenhagen (Other); Research Unit for General Practice in Aalborg (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, PROFESSOR, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APPI-MSK-OA-SELFIT
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis
Keywords: Exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-managed exercise (Experimental)
  Interventions: Behavioral: Self-managed exercise in a fitness center
- Physiotherapist-supervised exercise (Active Comparator)
  Interventions: Behavioral: Supervised Exercise

INTERVENTIONS:
Behavioral: Self-managed exercise in a fitness center — The participants are offered a 6-month membership of a local fitness club at no cost (paid by the trial). They will receive an introduction to the fitness centre and receive instructions from a personal trainer in the centre to create a personalized exercise programme
  Arms: Self-managed exercise
Behavioral: Supervised Exercise — The particiopants are offered participation in the usual care exercise delivered at municipal rehabilitation centers or private physiotherapy clinics, aat the discretion of the referring doctor.
  Arms: Physiotherapist-supervised exercise

SUMMARY:
Knee osteoarthritis (OA) is a common painful condition associated with pain and disability. OA healthcare costs the Danish society 4.6 billion DKK more per year than the non-OA population and we lack evidence on how best to organize and deliver care to reduce costs. Recommended first line treatment for knee OA is exercise with proven effects on symptoms. The current paradigm assumes that exercise needs to be delivered and supervised by a physiotherapist which require patients to attend a clinic at specific times and geographical locations. This is an expensive model of care and creates barriers for people that are active on the labor market or lives in remote areas with long distances to the nearest clinic. In fact, the productivity loss in Denmark associated with OA is estimated to be 12.4 billion DKK per year.

While effective on symptoms, the current model with supervised physiotherapy associates with significant shortcomings, and barriers related to patient heterogeneity, costs, accessibility, and work absenteeism.

As an alternative, a local fitness center is far more accessible as these are widely dispersed across the country, are accessible daily (including weekends) at all hours, is cheap and offers a wide variety of exercise types, classes, and equipment to accommodate individual preferences. The cost of a fitness center membership is approximately 300 DKK per month and includes exercise ad libitum. In contrast, a typical physiotherapist-supervised exercise program costs 3-4,000 DKK for a 2-month treatment with 2 weekly sessions.

Consequently, there is a need to investigate if self-managed exercise in a fitness center is cost-effective as first-line management of knee OA. To answer this question, the present trial aims to compare self-managed exercise in a fitness center to the current standard - supervised exercise. This has the potential to improve quality of care for people with knee OA by adding a cost-effective option for first line management of people with knee OA.

ELIGIBILITY:
Inclusion criteria

• Diagnosis of knee OA according to the NICE criteria: Adults aged 45 or over with activity-related joint pain and either no morning joint-related stiffness or morning stiffness that lasts no longer than 30 minutes.

Exclusion criteria

* Completion of a supervised therapeutic exercise program for knee OA within 3 months
* Contraindication to exercise (e.g., resting systolic blood pressure > 200 or diastolic blood pressure >110 mmHg, acute or reoccurring chest pain, unstable angina. uncontrolled cardiac arrhythmias, decompensated heart failure. suspected or known dissecting aortic aneurysm)
* Lack of independent mobility that requires aid for transportation to/from exercise facilities.
* Any condition or impairment that, in the opinion of the recruiting GP, makes a potential participant unsuitable for participation or which may obstruct participation (e.g. psychiatric or cognitive disorders, language barriers, or opiate dependency).

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain subscale of the KOOS (Knee injury and Osteoarthritis Outcome Score) questionnaire | Change from baseline after 3 months
  Assessed by the Knee injury and Osteoarthritis Outcome Score (KOOS) pain subscale (patient-reported questionnaire).
  The KOOS pain subscale consists of 9 questions with a five-point Likert scale scoring system (ranging from 0 (least severe) to 4 (most severe)). The answers are summed and a 0-100 normalized score is calculated with 0 indicating extreme pain and 100 indicating no pain.

SECONDARY OUTCOMES:
Health outcome and quality of life survey (EQ-5D-5L) | Change from baseline after 3 months
  EQ-5D-5L is a standardized patient-reported instrument for use as a measure of health outcome and quality of life. EQ-5D-5L is designed for self-completion by respondents and is ideally suited for use in surveys.
Patient Global Assessment of disease impact (PGA) | Change from baseline after 3 months
  Patient-reported degree of patient's perceived impact of their knee OA on their overall life will be obtained using a 100 mm analogue scale (VAS) with anchors: 0=" No impact" and 100 = "Worst imaginable impact".
KOOS Function subscale | Change from baseline after 3 months
  Assessed by the Knee injury and Osteoarthritis Outcome Score (KOOS) physical function subscale (patient-reported questionnaire). The KOOS physical function subscale consists of 17 questions with a five-point Likert scale scoring system (ranging from 0 (least severe) to 4 (most severe)). The answers are summed and a 0-100 normalized score is calculated with 0 indicating extreme functional impairment and 100 indicating no functional impairment.
KOOS quality of Life (QOL) subscale | Change from baseline after 3 months
  Assessed by the Knee injury and Osteoarthritis Outcome Score (KOOS) knee related quality of life subscale (patient-reported questionnaire) The KOOS knee related quality of life subscale consists of 4 questions with a five-point Likert scale scoring system (ranging from 0 (least severe) to 4 (most severe)). The answers are summed and a 0-100 normalized score is calculated with 0 indicating extremely poor knee related quality of life pain and 100 indicating very good knee related quality of life .
OMERACT-OARSI responder criteria | 3 months
  Number of treatment responders according to the OMERACT-OARSI response criteria. A participant is classified as a responder if at least 1of the following 2 conditions is observed:
  1. In either pain (KOOS pain subscale) or function (KOOS function subscale), a high improvement in the subscale, where high improvement in a subscale is achieved if there is both a >50% improvement from Baseline and an absolute change from Baseline of >20 points (0-100 scale), OR
  2. Improvement in at least two of the following three:
     * Improvement in pain (KOOS pain subscale) defined as >20% improvement from Baseline and an absolute change from Baseline of >10 points (0-100 scale).
     * Improvement in function (KOOS function subscale) defined as >20% improvement from Baseline and an absolute change from Baseline of > 10 points (0-100 scale).
     * Improvement in patient's global assessment defined as >20% improvement from Baseline and an absolute change from Baseline of >10 mm (0-100 scale).

OTHER OUTCOMES:
Analgesics usage | After 1, 2, 3, 4, 5, 6 months
  The participants' use of over-the-counter paracetamol and ibuprofen will be collected via questionnaire.
  Analgesics usage is recorded as a response to the questions "How often do you take pain relieving medicine* for your knee OA pain" with response options 1) Daily; 2) 2-3 times per week: 3) Rarer; or 4) Never. Responses 1 and 2 defines an analgesics user, whereas responses 3 and 4 defines a non-user.
  * A list of typical brand names will be provided.
Sleep Quality Single-item sleep quality scale (SQS) | After 1, 2, 3, 4, 5, 6 months
  Sleep quality will be obtained with the global Single-item sleep quality scale (SQS).
Self-reported physical activity (UCLA activity scale) | After 1, 2, 3, 4, 5, 6 months
  Self-reported physical activity will be obtained with the University of California Loas Angeles activity scale (UCLA). UCLA is a single-item 10-level-scale, ranging from level 10, representing a highly physically active patient, to level 1, a patient who is dependent on others and unable to leave home.
Out of pocket spending on knee OA - The cost for patients questionnaire (CoPaQ) | After 1, 2, 3, 4, 5, 6 months
  The cost for patients questionnaire (CoPaQ) is a comprehensive tool to measure direct and indirect out-of-pocket costs of a health condition for patients and their families to various outpatient contexts.
The World Health Organization Five Well-Being Index (WHO-5) | After 1, 2, 3, 4, 5, 6 months
  Self-reported mental well-being will be obtained with the WHO5-Well-Being Index consisting of five questions.
Body weight | After 1, 2, 3, 4, 5, 6 months
  Is recorded as kilograms and obtained self-reported via questionnaire
The KOOS (Knee injury and Osteoarthritis Outcome Score) questionnaire | After 1, 2, 3, 4, 5, 6 months
  The Knee injury and Osteoarthritis Outcome Score (KOOS) consists of 42 items covering five subscales (domains): 1) Pain; 2) Function; 3) Knee related quality of life; 4) Symptoms; 5) Sports and Recreation.
  The KOOS adopts a five-point Likert scale scoring system (ranging from 0 (least severe) to 4 (most severe)). A normalized score is calculated for each subscale (domain) with 100 indicating best score and 0 indicating the worst score.
Health outcome and quality of life survey (EQ-5D-5L) | After 1, 2, 4, 5, 6 months
  EQ-5D-5L is a standardized patient-reported instrument for use as a measure of health outcome and quality of life.
Patient Global Assessment of disease impact (PGA) | After 1, 2, 4, 5, 6 months
  Patient-reported degree of patient's perceived impact of their knee OA on their overall life will be obtained using a 100 mm analogue scale (VAS) with anchors: 0=" No impact" and 100 = "Worst imaginable impact".
OMERACT-OARSI responder criteria | After 6 months
  Number of treatment responders according to OMERACT-OARSI response criteria, following two conditions is observed at the post-baseline assessment:
  In either pain (KOOS pain subscale) or function (KOOS function subscale), a high improvement in the subscale, where high improvement in a subscale is achieved if there is both a > 50% improvement from Baseline and an absolute change from Baseline of > 20 points (0-100 scale), OR
  Improvement in at least two of the following three:
  Improvement in pain (KOOS pain subscale) defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 points (0-100 scale) Improvement in function (KOOS function subscale) defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 points (0-100 scale) Improvement in patient's global assessment defined as > 20% improvement from Baseline and an absolute change from Baseline of > 10 mm (0-100 scale)

IPD SHARING:
Plan to Share IPD: Yes
We will share the IPD, protocol and SAP, but the circumstances and timing has not been decided yet
Supporting Information: Study Protocol, SAP